CLINICAL TRIAL: NCT04254497
Title: A Comprehensive Evaluation of Circulating Tumor DNA and Circulating Tumor Cells as a Predictive Marker in Lung Cancer
Status: Completed | Type: Observational
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/216/B
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: EGFR mutation detection kit — A microsieve membrane filter device to effectively isolate circulating tumor cells from whole blood sample has been developed by the Institute of Bioengineering and Nanotechnology. The device exploits the size difference between cancer cells and blood cells to achieve the cancer cell capture on a microsieve filter with > 85% recovery rate from 4.5-ml whole blood within 10 min, demonstrated with cancer cells spiked into whole blood samples. The device contains a densely packed pore array (> 8000 pores/mm^2) with an optimized pore diameter of 10 µm. Fluid regulation and cell counting are achieved by a simple vacuum pumping and laboratory fluorescence microscope. The captured cells are stained with anti-EpCAM-PE for CTCs, anti-CD45-FITC for white blood cells, and 4',6-diamidino-2-phenylindole (DAPI) for cell nuclei. The CTCs are identified with anti-EpCAM positive, anti-CD45 negative and DAPI positive, characterized using a fluorescence microscope.

SUMMARY:
This study evaluates the use of ctDNA and CTCs in predicting disease activity and drug response in lung cancer patients and serves to complement existing methods to achieve a non-invasive and accurate means to guide treatment decisions.

DETAILED DESCRIPTION:
Lung cancer is not only amongst the top 3 most common cancer type in both men and women, but also the leading cause of cancer mortality in Singapore and the United States. Platinum-based chemotherapy is currently the mainstay in drug treatment for lung cancer patients although it only relieves disease-related symptoms temporarily. Recently, the use of molecularly targeted therapy has led to improved survival in subsets of patients. In particular, the presence of EGFR or ALK mutations from lung biopsies predicts improved response rate and progression-free survival from the use of tyrosine kinase inhibitors or crizotinib respectively. Importantly, EGFR mutations are more common in tumors of Asian patients (about 35%) versus non-Asians (about 10%).

The main cause of mortality in patients with solid cancers is metastases from dissemination via blood circulation. The ability to detect the presence of tumor cells in circulation even before overt metastases occur has evolved rapidly in recent years. The prognostic importance of circulating tumor DNA (ctDNA) and circulating tumor cells (CTCs) in several cancers has been found and this technique is widely recognized to be of major clinical and biologic importance. This study evaluates the use of ctDNA and CTCs in predicting disease activity and drug response in lung cancer patients and serves to complement existing methods to achieve a non-invasive and accurate means to guide treatment decisions.

Indeed, the use of ctDNA and CTCs as a marker for risk assessment and treatment monitoring is advantageous as it is accessible may be monitored on a regular basis on a non-invasive basis. This will better tailor our surveillance programmes and treatment to optimize disease outcomes.

The Investigators have developed an EGFR mutation detection kit that detects the 3 main EGFR mutations at ultrasensitive levels. The Investigators have applied this to a variety of clinical materials including formalin-fixed paraffin embedded DNA, pleural effusions, circulating DNA as well as circulating tumor cells and found that the kits can pick up these mutations with high sensitivity and specificity.

A microsieve membrane filter device to effectively isolate circulating tumor cells from whole blood sample has been developed by the Institute of Bioengineering and Nanotechnology. The device exploits the size difference between cancer cells and blood cells to achieve the cancer cell capture on a microsieve filter with > 85% recovery rate from 4.5-ml whole blood within 10 min, demonstrated with cancer cells spiked into whole blood samples. The device contains a densely packed pore array (> 8000 pores/mm^2) with an optimized pore diameter of 10 µm. Fluid regulation and cell counting are achieved by a simple vacuum pumping and laboratory fluorescence microscope. The captured cells are stained with anti-EpCAM-PE for CTCs, anti-CD45-FITC for white blood cells, and 4',6-diamidino-2-phenylindole (DAPI) for cell nuclei. The CTCs are identified with anti-EpCAM positive, anti-CD45 negative and DAPI positive, characterized using a fluorescence microscope.

Hence, from our preliminary studies, the investigators hypothesize that our technology is useful for isolating circulating tumour cells and that these circulating tumor cells likely correlate with disease activity and are not found in health individuals.

The monitoring of circulating tumor DNA and circulating tumour cells may provide a clinically valuable lead time in determining response, compared to conventional radiologic methods.

A cohort of patients will be recruited for a longitudinal cohort study where tissue and blood are collected for biomarkers. No intervention is envisioned. The study will be conducted over three years.

Patient Samples and Consent

Prospectively over six years(August 2014 to August 2020), about 150 patients diagnosed with lung cancer who provide full informed consent to this study will have tumor and/or blood and/or effusions collected. Patients from other locations may be referred to these sites.

If patients do not consent to collection of blood for clinical studies but have consented and signed informed operative consent for collection of frozen or formalin-fixed paraffin embedded material for research purposes including biopsies, cytology or surgical resections as part of the standard surgical consent form, tumor tissue and normal tissue will be collected from Changi General Hospital. Tumor staging and grading were obtained from review of the pathology reports and evaluation of the case notes by individual clinician investigators. Written informed consent for analysis of prospectively collected clinical samples will be obtained from all patients, including the consent to obtain a biopsy lung tissue specimen for research purpose. No other additional procedures are needed other than the recommended procedure to remove the patient's tissue for assessment of the tumour, be it bronchoscopy, CT-guided biopsy or open surgery, depending on physician's assessment. Once routine procedure is completed, one of the tissues will be selected for research purposes. The "research tissue blocks" will be anonymized and the slides batched for subsequent examination/verification of tumor presence by a pathologist.

Each prospective patient will provide baseline 3 EDTA tubes of blood (total approximately 30 ml). Urine (~100mL) will be collected at the same time for study of urine DNA.

These blood samples will be centrifuged for 10 minutes at 3000 rpm, for collection of serum and plasma for validation of biomarkers identified by microarray analysis, selecting for candidate secreted proteins in the blood.

Effusions (pleural or peritoneal) will be obtained as part of routine therapeutic procedures as recommended by the treating clinician, where the fluids would otherwise have been discarded. At no point will effusion fluid be obtained for the sole purpose of this study.

Downstream work in terms of evaluation of the CTCs, peripheral blood mononuclear cells, DNA, RNA, protein, and other genetic and molecular materials will be performed. Techniques applied will include quantitative PCR, sequencing, flow cytometry and immunophenotyping, immunohistochemistry, fluorescent in situ-hybridization, culture, etc.

Mutational analysis:

Genetic material will be extracted from 3-5 mL of materials trapped on sieve and from blood plasma, as well as relevant material such as effusions or urine. This will be analysed by quantitative PCR using custom designed primers and/or sequencing. Genetic materials will also be profiled using next-generation sequencing techniques to identify clinically actionable mutations such as BRAF, ALK, ROS, RET, etc.

Samples will be processed fresh. Any remaining sample will be separated into buffy coats and plasma and stored in liquid nitrogen and/or -80C.

Data and specimens are de-identified for laboratory processing. Each site will retain information linking patient to specimen. This is necessary for determination of follow-up.

Identified data will be located on a networked PC, physically located in Changi General Hospital and behind institutional firewalls. Individually identifiable data will be retained in the hospital and will not be shared with the laboratory.

The data will be archived for downstream projects once the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected to have lung cancer (determined by attending doctors).

Exclusion Criteria:

* None.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients (aged 21-99) suspected to have lung cancer will be recruited from Changi General Hospital. There are no restrictions based on the race of subject. We will exclude study participants who are unable to provide informed consent, such as children and mentally incapable individuals.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2014-09-11 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
Examine the sensitivity and specificity of our EGFR mutation detection kit in ctDNA, CTCs and matched tumor biopsies so as to examine their utility as a non-invasive liquid biopsy. | 6 years